CLINICAL TRIAL: NCT02033278
Title: Multicenter Phase IIb Clinical Trial, Double-blind, Randomized, Controlled Placebo for to Assess the Efficacy of Intracoronary Infusion of Autologous Adult Stem Cells Mononuclear Marrow Unexpanded on Functional Recovery in Patients With Idiopathic Dilated Cardiomyopathy and Heart Failure.
Brief Title: Infusion Intracoronary of Mononuclear Autologous Adult no Expanded Stem Cells of Bone Marrow on Functional Recovery in Patients With Idiopathic Dilated Cardiomyopathy and Heart Failure.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment rate, bibliographic evidence of lack of efficacy
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMMo/MD/2013
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Idiopathic Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusion of autologous mononuclear bone marrow cells (Experimental): Infusion of autologous mononuclear bone marrow cells plus conventional medical treatment (as indicated by clinician)
  Interventions: Drug: Infusion of autologous mononuclear bone marrow cells
- Placebo infusion (Placebo Comparator): Placebo infusion plus conventional medical treatment (as indicated by clinician)
  Interventions: Drug: Placebo infusion

INTERVENTIONS:
Drug: Infusion of autologous mononuclear bone marrow cells — Infusion of autologous mononuclear bone marrow cells plus conventional medical treatment (as indicated by clinician)
  Arms: Infusion of autologous mononuclear bone marrow cells
Drug: Placebo infusion — Placebo infusion plus conventional medical treatment (as indicated by clinician)
  Arms: Placebo infusion

SUMMARY:
Clinical trial phase IIb, double-blind, randomized, controlled with placebo. There is sufficient preliminary evidence to consider intracoronary injection of bone marrow progenitor cells as a viable, safe and beneficial treatment in patients with dilated cardiomyopathy, although the biological mechanism of action of bone marrow cells in the myocardium is not known. In this project we propose to investigate comparatively and from a biological and clinical point of view the applicability of regenerative therapy with autologous bone marrow cells in patients with dilated cardiomyopathy.

DETAILED DESCRIPTION:
The study population correspond to male and female patients with idiopathic dilated cardiomyopathy.

51 patients diagnosed with this disease are included. After inclusion, will proceed to the random allocation to study group or control group in a 2:1 ratio, 34 patients in the treatment group and 17 in the control group.

The total duration is expected to be 48 months: The inclusion period is 24 months and each patient assigned to the experimental group will be followed for 24 months, whereas that one ramdomized to the control group, will have a folow-up of 12 months. Upon completion there of, the patients will be followed in routine clinical practice.

This is a double blind study, in which all patients will perform the bone marrow harvesting.

All patients will receive the best medical treatment individualized (ACEIs or Angiotensin II receptor blocker, beta-blockers, diuretics and eplerenone) for at least 6 months prior to their participation in the clinical trial, so that the situation is stable and pharmacological basal condition is the same for everyone.

The bone marrow cells of patients assigned to placebo group will be cryopreserved, and once the trial is completed, the blind will be opened and all the patients who had been randomized to the control group, may be processed by the route of compassionate use with their own mononuclear bone marrow cells previously frozen.

The patients who are randomized to experimental group will be treated by the conventional treatment + infusion of autologous mononuclear bone marrow cells not expanded whereas the patients who are randomized to control group will be treated by the conventional treatment + infusion of placebo.

The main objective is to assess comparative the efficacy of intracoronary injection of bone marrow stem cells autologous to improve ventricular function in patients with idiopathic dilated cardiomyopathy who receive conventional medical treatment, compared with a control group who receive a infusion of placebo and conventional medical treatment. The improvement in ventricular function assessed by changes in angiographically determined ejection fraction.

Secondary objectives of the study are:

- To analyze the predictors of good clinical response, functional and biological treatment with adult stem cells autologous mononuclear bone marrow not expanded in terms of functional recovery.

The following parameters were evaluated: Functional class (NYHA), Natriuretic peptide B, Stress test (exercise time), Echocardiographic parameters of ventricular function, for example LVEF (%), TDV (ml), TSV (ml) and TAPSE (ms) and Biological parameters of cellular functionality, for example CD133 +, CD34 +, CD34 +/CD177 + and CD34 +/CD38- (in %).

- To determine, in the light of the obtained results, the application protocol suitable cell therapy for the treatment of dilated cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes and ages between 18 and 70 years.
2. Patients diagnosed with dilated cardiomyopathy established by echocardiography.
3. Minimum evolution since diagnosis of 6 months.
4. Absence of coronary injury tested with multislice CT and/or hemodynamic study performed after study entry, or within the previous 36 months (or before in specific low risk clinical profiles) if no angina symptomatology is present.
5. Patients receiving optimized medical therapy for at least 6 months prior to enrollment (individually adjusted according to functional status).
6. Ejection fraction of the left ventricle <40% or ejection fraction of the left ventricle 40% -50% if left ventricular tele-diastolic volume is > 110 ml/m2.
7. Presence of sinus rhythm.
8. Writen informed consent for participation in the trial.
9. Normal laboratory parameters, defined by: Leukocytes ≥ 3000; Neutrophils ≥ 1500; Platelets ≥ 100,000; Aspartate aminotransferase / Alanine aminotransferase ≤ 2.5 standard range institution; Creatinine ≤ 2.5 mg / dL; Haemoglobin > 9 g/dL
10. Women of childbearing potential must have negative results on a pregnancy test and agree to use medically approved methods of contraception thoughout follow up.

Exclusion Criteria:

1. Secondary Dilated cardiomyopathy.
2. Recent history of myocarditis (< 6 months prior to study entry).
3. Patients amenable to receive cardiac resynchronization therapy
4. Patients in active waiting list for heart transplantation.
5. Coexistence of other serious systemic diseases.
6. Coexistence of any type of blood disease
7. Pregnant or breastfeeding women; or women of childbearing potential not comminting to use effective contraception.
8. Patients who are currently participating, or have completed their participation in a clinical trial within the last 3 months. Patients who have participated in any advanced therapies clinical trial any time previously.
9. Patients with malignant or pre-malignant tumors.
10. Positive serology for hepatitis B virus, hepatitis C virus or human immunodeficiency virus.
11. Use of any protocolo prohibited medication. A wash-out period of 2 months can be considered for inclusion in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Changes in ventricular function measured angiographically. | 24 months

SECONDARY OUTCOMES:
Degree of clinical improvement based on the absence of major cardiac events (MACE) during follow-up. | 24 months
Clinical and analytical progress (NYHA grade & BNP) | 24 months
Time of evolution since diagnosis of idiopathic dilated cardiomyopathy prior to study entry. | 24 months
Functional recovery as measured with ergometry | 24 months
Echocardiography and Electrocardiography variables | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Romero Moreno, MD, PhD, Principal Investigator — Hospital Universitario Reina Sofía; Manuel Sobrino Marquez, MD, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Luis A Iñigo García, MD, Principal Investigator — Hospital Costa del Sol; Ricardo Zayas Rueda, MD, Principal Investigator — Hospital Universitario Puerta del Mar; Manuel De Mora Martín, MD, PhD, Principal Investigator — Hospital Regional U. Carlos Haya; Silvia López Fernández, MD, Principal Investigator — University Hospital Virgen de las Nieves; José Francisco Díaz Fernández, MD, Principal Investigator — Hospital Universitario Juan Ramón Jimenez; Jesús Oneto Otero, MD, Principal Investigator — Hospital de Jerez; Rafael Ruiz Salmerón, MD, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (9):
- Spain (9):
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hopistal Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Juan Ramón Jimenez, Huelva
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital Costa del Sol, Marbella
  - Hospital Regional U. Carlos Haya, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville

REFERENCES:
- [Derived] Romero M, Suarez-de-Lezo J, Herrera C, Pan M, Lopez-Aguilera J, Suarez-de-Lezo J Jr, Baeza-Garzon F, Hidalgo-Lesmes FJ, Fernandez-Lopez O, Martinez-Atienza J, Cebrian E, Martin-Palanco V, Jimenez-Moreno R, Gutierrez-Fernandez R, Nogueras S, Carmona MD, Ojeda S, Cuende N, Mata R. Randomised, double-blind, placebo-controlled clinical trial for evaluating the efficacy of intracoronary injection of autologous bone marrow mononuclear cells in the improvement of the ventricular function in patients with idiopathic dilated myocardiopathy: a study protocol. BMC Cardiovasc Disord. 2019 Aug 22;19(1):203. doi: 10.1186/s12872-019-1182-4. PMID 31438858